CLINICAL TRIAL: NCT06859749
Title: Does educatıonal Escape Game Affect Students' motıvatıon, academıc Self-effıcacy and Success Levels
Brief Title: Does educatıonal Escape Game Affect Students' motıvatıon, academıc Self-effıcacy and Success Levels: a quası-experımental Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: guzel
Record Dates: First submitted 2025-02-22; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Motivation; Self Efficacy
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Escape Game Group (Experimental): In order to perform the Escape game for students, 4 stations were prepared in the skills laboratory: "Pulse", "Respiration-Oxygen Saturation", "Blood Pressure", "Body Temperature". Separate scenarios will be prepared for each station.
  Interventions: Other: Education
- Question and Answer Group (No Intervention): Students will be given a question-answer application.

INTERVENTIONS:
Other: Education — Students will be given a question-answer application. In order to perform the Escape game for students, 4 stations were prepared in the skills laboratory: "Pulse", "Respiration-Oxygen Saturation", "Blood Pressure", "Body Temperature". Separate scenarios will be prepared for each station.
  Arms: Escape Game Group

SUMMARY:
This is a semi-experimental study. The study aimed to examine the effects of an educational escape game on students' motivation, academic self-efficacy and achievement levels. Students studying in an elderly care program will be included in the study. Students will be divided into 2 groups according to their branches: experimental (educational escape game) and control (question-answer).

H1. Students participating in the escape game will show significantly higher motivation in the "Motivation Scale for Teaching Materials" than students participating in the question-answer method.

H2. Students participating in the escape game will show significantly higher self-efficacy in the "Academic Self-Efficacy Scale" than students participating in the question-answer method.

H3. Students participating in the escape game will show significantly higher success in the "Achievement Test" than students participating in the question-answer method.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Receiving education in an elderly care program,
* Not having previously taken the "Elderly Care Principles and Practices I" and "Elderly Care Principles and Practices II" courses,
* Providing attendance during data collection processes.
* Having a phone and internet that can enter Google forms.

Exclusion Criteria:

* Being under 18 years of age,
* Not cooperating,
* Having previously taken the "Elderly Care Principles and Practices I" and "Elderly Care Principles and Practices II" courses,
* Being absent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Motivation average | 1 months
  The average scores of the students in the questionnaire used for motivation will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Muş Alparslan University, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will not be shared in order to ensure the privacy of the researchers.